CLINICAL TRIAL: NCT00001530
Title: Long-Term Results of DDD Pacing in Obstructive Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960059; 96-H-0059
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-04

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: Cardiac Hypertrophy; Drug-Refractory; Hemodynamic Benefits; Obstruction; Pacemaker Therapy; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomegaly; Bites and Stings

SUMMARY:
DDD pacing improves symptoms and relieves LV outflow tract (LVOT) obstruction in most patients with hypertrophic cardiomyopathy (HCM). Notably, when pacing is temporarily discontinued, the beneficial effects of pacing are evident in sinus rhythm. The long term results of this novel therapy are, however, uncertain. We propose (1) to record the hemodynamic changes following >4 years of pacing; and (2) to determine whether DDD pacing continues to be necessary in patients who have had a substantial relief of their LVOT obstruction. Patients who have had >50% reduction in LVOT pressure gradients will be randomized to two pacing modalities: DDD at 70 beats per minute and AAI pacing at 70 beats per minute (DDD switched off), and reevaluated after a six-month period.

DETAILED DESCRIPTION:
DDD pacing improves symptoms and relieves LV outflow tract (LVOT) obstruction in most patients with hypertrophic cardiomyopathy (HCM). Notably, when pacing is temporarily discontinued, the beneficial effects of pacing are evident in sinus rhythm. The long term results of this novel therapy are, however, uncertain. We propose (1) to record the hemodynamic changes following >4 years of pacing; and (2) to determine whether DDD pacing continues to be necessary in patients who have had a substantial relief of their LVOT obstruction. Patients who have had >50% reduction in LVOT pressure gradients will be randomized to two pacing modalities: DDD at 70 beats per minute and AAI pacing at 70 beats per minute (DDD switched off), and reevaluated after a six-month period.

ELIGIBILITY:
Group 1:

HCM patients, aged grater than 20 years of either gender who received DDD pacemakers at the NIH at least 4 years ago, for relief of LVOT obstruction and drug-refractory symptoms.

Group 2:

HCM patients selected from Group 1 who at the follow-up cardiac catheterization are demonstrated to have either (1) no significant LVOT obstruction (less than 30mm HG at rest and less than 50mm HG with Isuprel); or (2) a substantial reduction of the LVOT obstruction (greater than 50% reduction in LVOT gradient).

Patient who have developed a heart block will be excluded from group 2.

Females must have a negative pregnancy test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1996-04; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] McDonald K, McWilliams E, O'Keeffe B, Maurer B. Functional assessment of patients treated with permanent dual chamber pacing as a primary treatment for hypertrophic cardiomyopathy. Eur Heart J. 1988 Aug;9(8):893-8. doi: 10.1093/oxfordjournals.eurheartj.a062584. PMID 3181176
- [Background] Fananapazir L, Cannon RO 3rd, Tripodi D, Panza JA. Impact of dual-chamber permanent pacing in patients with obstructive hypertrophic cardiomyopathy with symptoms refractory to verapamil and beta-adrenergic blocker therapy. Circulation. 1992 Jun;85(6):2149-61. doi: 10.1161/01.cir.85.6.2149. PMID 1350522
- [Background] Fananapazir L, Epstein ND, Curiel RV, Panza JA, Tripodi D, McAreavey D. Long-term results of dual-chamber (DDD) pacing in obstructive hypertrophic cardiomyopathy. Evidence for progressive symptomatic and hemodynamic improvement and reduction of left ventricular hypertrophy. Circulation. 1994 Dec;90(6):2731-42. doi: 10.1161/01.cir.90.6.2731. PMID 7994815